CLINICAL TRIAL: NCT07272200
Title: Understanding Gene ENvironment Interaction in ALcohol-related Hepatocellular Carcinoma
Acronym: GENIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Serena Pelusi, Principal Investigator, Medical Doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Genial
Record Dates: First submitted 2025-02-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-02

CONDITIONS: HCC; Genetic Predisposition
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk factors (Experimental): In the context of the study, data will be collected to characterize clinical risk factors: biopsy parameters, lifestyle and metabolic factors (BMI, abdominal circumference (CA), smoking, alcohol, diet, ongoing medical therapy), liver fat content and liver damage (by abdominal ultrasound and Fibroscan measurement of liver stiffness, liver stiffness measurement (LSM) and controlled attenuation parameter (CAP)).
  Interventions: Other: quantify of risk factors

INTERVENTIONS:
Other: quantify of risk factors — the impact of risk factors and their interaction on the incidence of disease through a score that predicts HCC and select patients for whom screening is convenient.

SUMMARY:
It has been estimated that alcohol causes around 40% of premature liver deaths in Europe each year, although this number is probably underestimated. Alcohol-related liver disease (ALD) is the most common cause of liver cirrhosis and liver death in Europe with a peak age of deaths occurring among individuals aged 40 to 50. Despite these findings, ALD is little studied with only 5% of all clinical trials in the field of liver disease recorded on ClinicalTrials.gov and only 5% of all publications in the same research area.

Liver cancer is the second most common cause of cancer-related death (15-20% survival at 5 years) and the second most common cause of alcohol-related cancers worldwide.

Like other complex diseases, ALD-HCC results from the interaction between environmental determinants and genetic variations but knowledge of gene-environment interactions is currently lacking in this area. The GENIAL project will address these needs through a comprehensive evaluation of gene-environment interactions concerning ALD-HCC.

ELIGIBILITY:
Inclusion Criteria:

Patients from the EPIDEMIC (approval no. 1822 of 27 August 2013) and SERENA (last amendment no. 1151_2021 of 9 November 2021), already approved by the CE Milano Area 2 will be included.

* Diagnosis of NAFLD or cryptogenic liver disease, allowing a more liberal alcohol intake limit (<60/40 g/day in M/F), so that subjects with a moderate alcoholic component of the hepatopathy are also included, Important factor given the high epidemiological weight of this group
* Any of the following:
* Male patient with type 2 diabetes or obesity carrying at least three genetic variants in PNPLA3, TM6SF2, MBOAT7.
* Willingness to sign informed consent.

Exclusion Criteria:

* Alcohol intake >60/40 g/day in M/F
* Chronic viral or autoimmune hepatitis
* Any previously diagnosed liver genetic disease associated with increased risk of HCC (such as hereditary hemochromatosis, Wilson's disease, Alpha-1 antitrypsin deficiency)
* Use of drugs known to induce steatosis and liver disease
* HCC previously diagnosed the study start date.
* Other pathological conditions with prognosis less than two years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of genetic risk factors | up to 60 months
  The research aims to conduct the Measurement of the Frequency/Incidence (expressed as the percentage of the study population) of new genetic variants, identified using DNA Sequencing and subsequent bioinformatics analysis, that are associated with HCC in patients with ALD and related NAFLD. This measurement will be followed by the assessment of the CORRELATION between the newly identified genetic variants and the Prevalence (expressed as the percentage of the general population) of the clinical phenotype ALD-HCC.

SECONDARY OUTCOMES:
Impact of genetic risk factor | up to 60 months
  The primary goal is the assessment of the Predictive Capacity (measured via Area Under the Receiver Operating Characteristic Curve (AUC) and P-value) of a newly created Polygenic-Clinical Risk Score (PRS-C) for the development of HCC. Subsequently, the Predictive Accuracy (measured in percentage of correct predictions, Sensitivity, and Specificity) of an Artificial Intelligence (AI) Algorithm will be evaluated. This Algorithm will be trained by integrating the aforementioned PRS (derived from the combination of genetic and non-genetic information) and other clinical and demographic variables, aiming to obtain predictive information on the individual risk of developing the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT07272200/Prot_SAP_000.pdf